CLINICAL TRIAL: NCT00571142
Title: Pars Plana Vitrectomy and Bevacizumab for the Treatment of Diffuse Diabetic Macular Edema (A Pilot Study)
Brief Title: Vitrectomy and Bevacizumab for Diffuse Diabetic Macular Edema
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Veronica Kon-Jara MD, Asociacion para Evitar la Ceguera en Mexico I.A.P.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC-ret
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Diffuse Diabetic Macular Edema
Keywords: edema; retinal thickness; diabetic retinopathy
MeSH Terms: conditions — Edema; Diabetic Retinopathy | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Renal disease
  Interventions: Procedure: Bevacizumab + Pars plana vitrectomy
- 2 (Active Comparator): Without renal disease
  Interventions: Procedure: Bevacizumab + pars plana vitrectomy

INTERVENTIONS:
Procedure: Bevacizumab + Pars plana vitrectomy — 2.5 mg / 0.1 ml bevacizumab after pars plana vitrectomy. Limitorexis would be optional.
  Arms: 1
Procedure: Bevacizumab + pars plana vitrectomy — 2.5 mg /0.1 ml of bevacizumab after pars plana vitrectomy
  Arms: 2

SUMMARY:
To Evaluate combined effect of vitrectomy and bevacizumab to stabilize retinal thickness and visual acuity in patients with diffuse diabetic macular edema and their relation to renal disease.

ELIGIBILITY:
Inclusion Criteria:

* Older than 25 yo
* Diffuse diabetic macular edema with or without previous treatment

Exclusion Criteria:

* Another retinal disease
* Pregnancy

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2007-11 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Retinal thickness | 3 months

SECONDARY OUTCOMES:
Visual acuity | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Kon-Jara, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociacion para Evitar la Ceguera en Mexico I.A.P., México, Mexico